CLINICAL TRIAL: NCT00862251
Title: A Randomized, Double-Blind, Active-Controlled Study of Patients With Cardiovascular Disease and Diabetes Mellitus Not Adequately Controlled With Simvastatin or Atorvastatin: Comparison of Switching to Combination Tablet Ezetimibe/Simvastatin Versus Switching to Rosuvastatin or Doubling the Statin Dose
Brief Title: Ezetimibe/Simvastatin (MK-0653A) Versus Rosuvastatin Versus Doubling Statin Dose in Participants With Cardiovascular Disease and Diabetes Mellitus (MK-0653A-133)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-133; 2009_559 (Other: Merck Study Number)
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Disorder; Diabetes Mellitus
Keywords: cardiovascular disorder
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus | interventions — Ezetimibe, Simvastatin Drug Combination; Simvastatin; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ezetimibe/simvastatin (Experimental)
  Interventions: Drug: ezetimibe (+) simvastatin; Drug: atorvastatin 10 mg or simvastatin 20 mg
- Doubling statin dose (Active Comparator)
  Interventions: Drug: simvastatin 40 mg or atorvastatin 20 mg; Drug: atorvastatin 10 mg or simvastatin 20 mg
- Rosuvastatin (Active Comparator)
  Interventions: Drug: Rosuvastatin; Drug: atorvastatin 10 mg or simvastatin 20 mg

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — ezetimibe/simvastatin 10/20 mg tablets, taken once daily for six weeks.
  Other Names: Vytorin
  Arms: Ezetimibe/simvastatin
Drug: simvastatin 40 mg or atorvastatin 20 mg — simvastatin 40 mg or atorvastatin 20 mg tablets, taken once daily for six weeks.
  Other Names: Lipitor, Zocor
  Arms: Doubling statin dose
Drug: Rosuvastatin — rosuvastatin 10 mg tablets, taken once daily for six weeks.
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: atorvastatin 10 mg or simvastatin 20 mg — All patients will take atorvastatin 10 mg tablets OR simvastatin 20 mg tablets, taken once daily in a 6-week screening/stabilization period prior to randomization.
  Other Names: Lipitor, Zocor

SUMMARY:
The purpose of this study is to determine the efficacy of switching to a combination tablet ezetimibe/simvastatin (10mg/20mg) versus rosuvastatin (10 mg) versus doubling the statin dose in those patients who have cardiovascular disease and diabetes mellitus not adequately controlled on simvastatin 20 mg or atorvastatin 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patient has not taken common statins or ezetimibe within 6 weeks of study screening or patient is currently taking a daily dose of the following statins for 6 weeks prior to study screening: simvastatin, atorvastatin, pravastatin, fluvastatin, ezetimibe, lovastatin, or ezetimibe + fluvastatin
* Patient is willing to go on a cholesterol and glucose lowering diet for the duration of the study
* Patient is willing to remain abstinent or use birth control for the duration of the study
* Patient has Diabetes Mellitus with cardiovascular disease

Exclusion Criteria:

* Patient has sensitivity to certain common statin drugs
* Patient is Asian and would not be able to start taking the higher doses of rosuvastatin necessary for the study design
* Patient consumes more than 2 alcoholic drinks per day
* Patient is pregnant or breast-feeding
* Patient has been treated with other investigational drugs within 30 days of first visit
* Patient is currently on prohibited doses of the following statin drugs: rosuvastatin, simvastatin, atorvastatin, and pravastatin
* Patient has congestive heart failure
* Patient has uncontrolled high blood pressure
* Patient has kidney disease
* Patient has uncontrolled endocrine or metabolic disease which are known to possibly increase blood lipoproteins
* Patient has diabetes mellitus that is not well controlled
* Patient is human immunodeficiency virus (HIV) positive
* Patient is currently taking medications that inhibit Cytochrome P450 3A4 (CYP3A4)
* Patient is currently taking therapies that would increase the risk of muscle weakness
* Patient has been taking certain over- the-counter lipid-lowering agents within 6 weeks prior to visit 1
* Patient is currently taking psyllium or other fiber-based laxatives

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le NA, Tomassini JE, Tershakovec AM, Neff DR, Wilson PW. Effect of Switching From Statin Monotherapy to Ezetimibe/Simvastatin Combination Therapy Compared With Other Intensified Lipid-Lowering Strategies on Lipoprotein Subclasses in Diabetic Patients With Symptomatic Cardiovascular Disease. J Am Heart Assoc. 2015 Oct 20;4(10):e001675. doi: 10.1161/JAHA.114.001675. PMID 26486166
- [Derived] Rosen JB, Jimenez JG, Pirags V, Vides H, Massaad R, Hanson ME, Brudi P, Triscari J. Consistency of effect of ezetimibe/simvastatin compared with intensified lipid-lowering treatment strategies in obese and non-obese diabetic subjects. Lipids Health Dis. 2013 Jul 16;12:103. doi: 10.1186/1476-511X-12-103. PMID 23866306
- [Derived] Rosen JB, Jimenez JG, Pirags V, Vides H, Hanson ME, Massaad R, McPeters G, Brudi P, Triscari J. A comparison of efficacy and safety of an ezetimibe/simvastatin combination compared with other intensified lipid-lowering treatment strategies in diabetic patients with symptomatic cardiovascular disease. Diab Vasc Dis Res. 2013 May;10(3):277-86. doi: 10.1177/1479164112465212. Epub 2013 Jan 3. PMID 23288881
- [Derived] Jimenez JG, Rosen JB, Pirags V, Massaad R, Hanson ME, Brudi P, Triscari J. The efficacy and safety of ezetimibe/simvastatin combination compared with intensified lipid-lowering treatment strategies in diabetic subjects with and without metabolic syndrome. Diabetes Obes Metab. 2013 Jun;15(6):513-22. doi: 10.1111/dom.12059. Epub 2013 Jan 25. PMID 23279632

RESULTS

PARTICIPANT FLOW:
Groups:
- Ezetimibe/Simvastatin: Ezetimibe/simvastatin 10/20 mg tablets, taken once daily for six weeks
- Doubling Statin Dose: simvastatin 40 mg or atorvastatin 20 mg tablets, taken once daily for six weeks.
Period: Overall Study
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Started | 322 | 162 | 324
Completed | 303 | 157 | 315
Not Completed | 19 | 5 | 9
Not completed — Adverse Event | 8 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 1
Not completed — Withdrawal by Subject | 9 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin | Total
Number analyzed (Participants) | 322 | 162 | 324 | 808
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.8) | 64.7 (8.3) | 63.6 (8.4) | 64.0 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 82 | 142 | 386
  Male | 160 | 80 | 182 | 422

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) After Switching to Treatment With Ezetimibe/Simvastatin vs Doubling the Dose of Statin (Simvastatin or Atorvastatin).
Time Frame: Baseline and Week 6
Population: Efficacy data were analyzed using the full analysis set (FAS) population defined as all randomized participants who received at least one dose of blinded study treatment and had baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose
Number analyzed (Participants) | 314 | 159
Percent change | -23.13 [-25.95 to -20.31] | -8.37 [-12.32 to -4.41]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis (LDA); Percent change in least-square means = -14.76, 95% CI 2-sided [-19.61 to -9.91]

2. Secondary Outcome: In Participants Treated With Simvastatin at Baseline, Percent Change From Baseline in LDL-C After Switching to Treatment With Ezetimibe/Simvastatin vs Doubling the Dose of Simvastatin
Time Frame: Baseline and Week 6
Population: Analysis performed on subpopulation of participants who were previously treated with simvastatin 20 mg and were switched to either Ezetimibe/simvastatin or had simvastatin dose doubled to 40 mg
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Doubling Simvastatin Dose: simvastatin 40 mg tablets, taken once daily for six weeks.
Arm/Group | Ezetimibe/Simvastatin | Doubling Simvastatin Dose
Number analyzed (Participants) | 158 | 78
Percent change | -21.59 [-25.54 to -17.65] | -7.98 [-13.57 to -2.38]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Simvastatin Dose; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis (LDA); Percent change in Least Square Means = -13.62, 95% CI 2-sided [-20.44 to -6.79]

3. Secondary Outcome: In Participants Treated With Atorvastatin at Baseline, Percent Change From Baseline in LDL-C After Switching to Treatment With Ezetimibe/Simvastatin vs Doubling the Dose of Atorvastatin
Time Frame: Baseline and Week 6
Population: Analysis performed on subpopulation of participants who were previously treated with atorvastatin 10 mg and were switched to either Ezetimibe/simvastatin or had atorvastatin dose doubled to 20 mg
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Doubling Atorvastatin Dose: atorvastatin 20 mg tablets, taken once daily for six weeks.
Arm/Group | Ezetimibe/Simvastatin | Doubling Atorvastatin Dose
Number analyzed (Participants) | 156 | 81
Percent change | -24.58 [-28.63 to -20.53] | -8.85 [-14.47 to -3.23]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Atorvastatin Dose; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis (LDA); Percent change in least squares mean = -15.73, 95% CI 2-sided [-22.65 to -8.81]

4. Secondary Outcome: Percent Change From Baseline in LDL-C After Switching to Treatment With Ezetimibe/Simvastatin vs Switching Treatment to Rosuvastatin
Time Frame: Baseline and Week 6
Population: Efficacy data were analyzed primarily based upon the full analysis set (FAS) population defined as all randomized participants who received at least one dose of blinded study treatment and had baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Rosuvastatin
Number analyzed (Participants) | 314 | 315
Percent change | -23.13 [-25.95 to -20.31] | -19.32 [-22.14 to -16.51]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.060, Longitudinal Data Analysis; Percent Change in Least Squares Means = -3.81, 95% CI 2-sided [-7.78 to 0.17]

5. Secondary Outcome: Number of Participants Who Reached the Target LDL-Cholesterol Level of < 70 mg/dL (1.81 mmol/L)
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 314 | 159 | 315
participants | 171 | 43 | 134
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.9, 95% CI 2-sided [2.5 to 6.2]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.3 to 2.6]

6. Secondary Outcome: In Participants Treated With Simvastatin at Baseline, Number of Participants Who Reached the Target LDL-Cholesterol Level of < 70 mg/dL (1.81 mmol/L)
Time Frame: Week 6
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Ezetimibe/Simvastatin | Doubling Simvastatin Dose
Number analyzed (Participants) | 158 | 78
participants | 84 | 19
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Simvastatin Dose; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.5, 95% CI 2-sided [2.3 to 8.5]

7. Secondary Outcome: In Participants Treated With Atorvastatin at Baseline, Number of Participants Who Reached the Target LDL-Cholesterol Level of < 70 mg/dL (1.81 mmol/L)
Time Frame: Week 6
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Ezetimibe/Simvastatin | Doubling Atorvastatin Dose
Number analyzed (Participants) | 156 | 81
participants | 87 | 24
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Atorvastatin Dose; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.5, 95% CI 2-sided [1.9 to 6.6]

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC)
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 314 | 159 | 315
Percent Change | -13.21 (17.69) [-14.99 to -11.43] | -4.88 (15.14) [-7.37 to -2.39] | -10.58 (15.18) [-12.36 to -8.81]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis (LDA); Least Squares Mean Difference = -8.33, 95% CI 2-sided [-11.38 to -5.28]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.039, Longitudinal data analysis (LDA); Least Squares Mean Difference = -2.63, 95% CI 2-sided [-5.13 to -0.13]

9. Secondary Outcome: Percent Change From Baseline in Triglycerides
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 314 | 159 | 315
Percent change | -5.51 [-8.75 to -2.15] | -2.63 [-7.23 to 2.21] | -3.35 [-6.66 to 0.08]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p = 0.316, Longitudinal data analysis (LDA); Least Squares Mean Difference = -2.88, 95% CI 2-sided [-8.53 to 2.77]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.356, Longitudinal data analysis (LDA); Least Squares Mean Difference = -2.16, 95% CI 2-sided [-6.75 to 2.43]

10. Secondary Outcome: Percent Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C)
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 314 | 159 | 315
percent change | 1.47 [-0.27 to 3.21] | 1.00 [-1.43 to 3.43] | 1.99 [0.26 to 3.73]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p = 0.756, Longitudinal data analysis (LDA); Least Squares Mean Difference = 0.47, 95% CI 2-sided [-2.50 to 3.45]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.675, Longitudinal data analysis (LDA); Least Sqares Mean Difference = -0.52, 95% CI 2-sided [-2.96 to 1.92]

11. Secondary Outcome: Percent Change From Baseline in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 314 | 159 | 315
Percent change | -18.39 [-20.90 to -15.88] | -6.77 [-10.29 to -3.25] | -15.14 [-17.72 to -12.70]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis (LDA); Least Squares Mean Difference = -11.62, 95% CI 2-sided [-15.93 to -7.31]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.078, Longitudinal data analysis (LDA); Least Squares Mean Difference = -3.18, 95% CI 2-sided [-6.71 to 0.35]

12. Secondary Outcome: Percent Change From Baseline in LDL-C/HDL-C Ratio
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 314 | 159 | 315
Percent change | -21.55 [-25.09 to -18.01] | -7.39 [-12.34 to -2.43] | -18.99 [-22.52 to -15.46]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis (LDA); Least Squares Mean Difference = -14.16, 95% CI 2-sided [-20.23 to -8.10]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.313, Longitudinal data analysis (LDA); Least Sqares Mean Difference = -2.56, 95% CI 2-sided [-7.53 to 2.41]

13. Secondary Outcome: Percent Change From Baseline in TC/HDL-C Ratio
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 314 | 159 | 315
Percent change | -12.52 [-14.83 to -10.22] | -4.36 [-7.58 to -1.14] | -10.70 [-12.99 to -8.40]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis (LDA); Least Squares Mean Difference = -8.17, 95% CI 2-sided [-12.10 to -4.23]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.266, Longitudinal data analysis (LDA); Least Squares Mean Difference = -1.83, 95% CI 2-sided [-5.05 to 1.40]

14. Secondary Outcome: Percent Change From Baseline in Non-HDL-C/HDL-C Ratio
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 314 | 159 | 315
percent change | -16.77 [-20.09 to -13.45] | -5.32 [-9.98 to -0.66] | -14.64 [-17.95 to -11.32]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis (LDA); Least Squares Mean Difference = -11.45, 95% CI 2-sided [-17.16 to -5.75]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.371, Longitudinal data analysis (LDA); Least Squares Mean Difference = -2.13, 95% CI 2-sided [-6.81 to 2.54]

15. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B)
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 313 | 159 | 313
Percent change | -14.98 [-16.99 to -12.97] | -6.97 [-9.78 to -4.15] | -12.03 [-14.05 to -10.02]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis (LDA); Least Squares Mean Difference = -8.01, 95% CI 2-sided [-11.46 to -4.56]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.041, Longitudinal data analysis (LDA); Least Squares Mean Difference = -2.95, 95% CI 2-sided [-5.78 to -0.12]

16. Secondary Outcome: Percent Change From Baseline Apolipoprotein A-I (Apo A-I)
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 313 | 159 | 313
Percent change | 0.64 [-0.84 to 2.11] | -0.93 [-2.99 to 1.12] | 0.86 [-0.62 to 2.34]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p = 0.218, Longitudinal data analysis (LDA); Least Squares Mean Difference = 1.57, 95% CI 2-sided [-0.93 to 4.06]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.832, Longitudinal data analysis (LDA); Least Squares Mean Difference = -0.22, 95% CI 2-sided [-2.27 to 1.83]

17. Secondary Outcome: Percent Change From Baseline in Apo B/Apo A-I Ratio
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 313 | 159 | 313
Percent change | -13.67 [-16.27 to -11.06] | -4.75 [-8.39 to -1.11] | -11.14 [-13.75 to -8.54]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis (LDA); Least Squares Mean Difference = -8.91, 95% CI 2-sided [-13.36 to -4.47]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.175, Longitudinal data analysis (LDA); Least Squares Mean Difference = -2.52, 95% CI 2-sided [-6.17 to 1.13]

18. Secondary Outcome: Percent Change From Baseline in High-sensitivity C-reactive Protein (Hs-CRP)
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Number analyzed (Participants) | 313 | 159 | 315
Percent change | -4.42 [-13.94 to 6.15] | -1.64 [-14.93 to 13.74] | -9.11 [-18.13 to 0.92]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Doubling Statin Dose; Test type: Superiority or Other; p = 0.749, Longitudinal data analysis (LDA); Least Squares Mean Difference = -2.78, 95% CI 2-sided [-19.88 to 14.32]
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.494, Longitudinal data analysis (LDA); Least Squares Mean Difference = 4.69, 95% CI 2-sided [-8.73 to 18.10]

ADVERSE EVENTS:
Description: All Patients as Treated (APaT) population was used for the analysis of safety data. The APaT population consisted of all randomized patients who received at
  least one dose of study treatment.
Arm/Group | Ezetimibe/Simvastatin | Doubling Statin Dose | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 2/321 | 1/162 | 2/323
Other Adverse Events (participants affected / at risk) | 0/321 | 0/162 | 0/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe/Simvastatin (N=321) | Doubling Statin Dose (N=162) | Rosuvastatin (N=323)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An investigator and/or his/her colleagues may publish the results for their study site independently after the multicenter publication, or 24 months after completion of the study, whichever comes first. The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.